CLINICAL TRIAL: NCT05169723
Title: Respiratory Emissions in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CIA-292
Record Dates: First submitted 2021-12-08; First posted 2021-12-27 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Respiratory Activity 1 (Experimental)
  Interventions: Behavioral: Exertional respiratory activities
- Respiratory Activity 2 (Experimental)
  Interventions: Behavioral: Exertional respiratory activities
- Respiratory Activity 3 (Experimental)
  Interventions: Behavioral: Exertional respiratory activities

INTERVENTIONS:
Behavioral: Exertional respiratory activities — participants will perform a series of exertional respiratory activities

SUMMARY:
This is an randomised cross over trial in healthy participants measuring respiratory emissions during different respiratory activities.

ELIGIBILITY:
Inclusion Criteria:

* Adults, over the age of 18 and able to give informed consent
* Symptom free from any respiratory illness in the last 48 hours

Exclusion Criteria:

* Pregnant (where the participant feels that their pregnancy will make participation uncomfortable)
* Inability to give consent
* Current respiratory disease. Participants with well controlled asthma will be included (defined as asthma that the participant self-rates their asthma as being under control and that does not limit exercise, work)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Count of total number of respiratory particles emitted during respiratory activities in the range of 0.3 to 25 microns | Emission of particles will be collected and analysed for 2 minutes during each experimental condition
  Particles emitted will be counted using two different optical particle counters

CONTACTS AND LOCATIONS:
Locations (1):
- Fisher and Paykel Healthcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No